CLINICAL TRIAL: NCT01670500
Title: A Randomized Phase II Trial of Neoadjuvant Cisplatin vs. Doxorubicin/Cyclophosphamide (AC) in Women With Newly Diagnosed Breast Cancer and Germline BrCa Mutations
Brief Title: Cisplatin vs. Doxorubicin/Cyclophosphamide in BrCa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nadine Tung, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-258
Record Dates: First submitted 2012-08-16; First posted 2012-08-22 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: germline mutation; BRCA1 mutation; BRCA2 mutation
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxorubicin-Cyclophosphamide (Active Comparator): Doxorubicin q 2-3 wk x 4 Cyclophosphamide q 2-3 wk x 4
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin
- Cisplatin (Active Comparator): Cisplatin q 3 wk x 4
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — administered intravenously every 3 weeks for 4 doses
  Other Names: cisplatinum, or cis-diamminedichloroplatinum(II) (CDDP)
  Arms: Cisplatin
Drug: Cyclophosphamide — administered with doxorubicin intravenously every 2 or 3 weeks for 4 doses
  Other Names: Cytoxan
  Arms: Doxorubicin-Cyclophosphamide
Drug: Doxorubicin — administered with Cyclophosphamide intravenously every 2 or 3 weeks for 4 doses
  Other Names: Adriamycin
  Arms: Doxorubicin-Cyclophosphamide

SUMMARY:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational drug, which is cisplatin in this trial, to learn how well it works in treating a specific cancer. "Investigational" means that cisplatin is still being studied for use in this setting and that research doctors are trying to find out more about it-in this case, how effective cisplatin is for treating breast cancer in BRCA mutation carriers. It also means that the FDA has not yet approved cisplatin for your type of cancer. Cisplatin has been approved by the FDA for treatment of other cancers.

The purpose of this study is to evaluate cisplatin, a chemotherapy drug that has been shown to be active in the treatment of women with breast cancer and a BRCA mutation. In this study, we are comparing cisplatin to the standard chemotherapy, doxorubicin and cyclophosphamide ("AC") that you might receive if you did not participate in this study.

DETAILED DESCRIPTION:
If screening tests show that you are eligible to participate in the research study you will begin study treatment. You may undergo an optional research biopsy so the study team can obtain tissue samples. This will be used for biomarker research and will help your doctors to better understand your disease, how the drug is working in your body, and may help to identify which people may benefit most from platinum or from adriamycin/cytoxan in the future.

Because no one knows which of the study options is best, you will be "randomized" to receive either cisplatin or doxorubicin and cyclophosphamide ("AC") chemotherapy prior to removal of your breast cancer. Chemotherapy administered before the removal of the cancer is known as neoadjuvant chemotherapy. Randomization means that you are put into a group by chance. It is like flipping a coin. Neither you nor the research doctor will choose what group you will be in. You will have an equal chance of being placed in either group.

If you are randomized to receive cisplatin you will receive cisplatin once every three weeks for a total of four doses. You will be given cisplatin by vein (IV) on the first day of each treatment cycle. The cisplatin infusion can take between 1 to 2 hours. Before and after receiving cisplatin, you will receive fluid hydration by vein, and you will also be given medicine to help prevent side effects such as nausea. The total time of the infusion of cisplatin and the additional fluid and medications will take about 6 hours. After you receive cisplatin, you will be asked to drink about 12 eight ounce glasses of fluid per day, especially 2 or 3 days after therapy. The study treatment will stop if you have serious side effects or if the tumor grows despite receiving cisplatin chemotherapy.

If you are randomized to "AC" chemotherapy you will receive both doxorubicin and cyclophosphamide once every 2 or 3 weeks for a total of four doses by vein on the first day of each treatment cycle. The interval between chemotherapy will be decided by your research doctor. If you receive the chemotherapy every two weeks, you will also receive a subcutaneous injection the day after chemotherapy. This injection contains a medicine that contains a growth factor that will boost your immune system in order to allow your body to be ready for chemotherapy in two weeks. The study treatment will be stopped if you have serious side effects or if the tumor grows despite the doxorubicin and cyclophosphamide chemotherapy.

At the beginning of each treatment cycle you will have a physical exam (including weight and vital signs) and you will be asked general questions about your health and any medications you may be taking, as well as specific questions about any side effects you may be experiencing while receiving study treatment. Prior to each cycle of chemotherapy, you will have standard blood tests to check your blood counts. If you are receiving cisplatin your kidney function and body salts will also be checked prior to each chemotherapy cycle. In addition, 7-10 days after chemotherapy your blood will be drawn to look at your blood cell count to determine your risk of infection; if you have received cisplatin, your kidney function and blood electrolytes will also be evaluated. The blood draw performed 7-10 days after chemotherapy can be done in the hospital where you received your chemotherapy or closer to home. About 1 tablespoon of blood will be drawn for these tests.

Surgery to remove your tumor will occur within six weeks after the last dose of chemotherapy. Your surgery will be performed by your surgeon, as part of the standard care for your disease.

Your treating physician or nurse practitioner will examine you to assess your tumor each time you receive chemotherapy. A measurement of your tumor will be performed on the first day of each treatment cycle as part of your physical exam. After the slides of your initial breast cancer biopsy have been reviewed at your hospital, these slides and your tumor block will be sent to the study pathologist at DF/HCC. Likewise, after chemotherapy, your breast cancer will be removed by lumpectomy or mastectomy. After these slides are reviewed at your hospital, they will also be sent with the tumor block to the study pathologist so that the response of your tumor to the study treatment can be assessed. After these slides are reviewed, they will be returned to the hospital at which the biopsy and surgery were performed.

Decisions about whether you will receive more chemotherapy after your surgery is up to your treating physicians. If you receive chemotherapy, the choice of chemotherapy is also up to your doctors. Decisions about post-operative chemotherapy are not part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of invasive breast cancer
* Stage: Clinical T1 >/= 1.0 cm, T2 or T3, N0-3, M0
* HER2 negative
* ER and PgR status by immunohistochemistry must be known. ER positive patients are allowed if physicain has determined neoadjuvant chemo is appropriate.
* Life expectancy greater than six months
* Use of an effective means of contraception is required

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior anthracycline or platinum based therapy
* Prior treatment for the current breast cancer, including chemotherapy, hormonal therapy, radiation or experimental therapy
* Ipsilateral breast recurrence, unless prior treatment consisted of excision alone for DCIS or breast-conserving treatment and hormonal therapy for DCIS or invasive cancer
* Peripheral neuropathy of any etiology that exceeds grade 1
* Significant hearing loss
* Renal dysfunction
* Use of other investigational or study agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs
* Uncontrolled intercurrent illness
* Any condition that would prohibit administration of corticosteroids
* Uncontrolled diabetes
* Pre-existing medical condition that would represent toxicity in excess of grade 1 as measured by CTCAE (unless not considered medically significant by the physician)
* Known HIV positive individuals on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-10; Primary Completion 2019-05 (Actual); Study Completion 2025-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Tung, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (15):
- United States (15):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Smilow Cancer Hospital Care Center at Derby, Derby, Connecticut
  - Smilow Cancer Hospital Care Center at Guilford, Guilford, Connecticut
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University, Durham, North Carolina
  - Women and Infants Hospital, Providence, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Takamizawa S, Ishiki H, Shimoi T, Shimizu M, Satomi E. Neoadjuvant Cisplatin in BRCA Carriers With HER2-Negative Breast Cancer. J Clin Oncol. 2020 Aug 10;38(23):2699-2700. doi: 10.1200/JCO.20.00789. Epub 2020 Jun 9. No abstract available. PMID 32516091
- [Derived] Tung N, Hacker MR, Garber JE. Reply to S. Takamizawa et al. J Clin Oncol. 2020 Aug 10;38(23):2700-2701. doi: 10.1200/JCO.20.01190. Epub 2020 Jun 9. No abstract available. PMID 32516090
- [Derived] Tung N, Arun B, Hacker MR, Hofstatter E, Toppmeyer DL, Isakoff SJ, Borges V, Legare RD, Isaacs C, Wolff AC, Marcom PK, Mayer EL, Lange PB, Goss AJ, Jenkins C, Krop IE, Winer EP, Schnitt SJ, Garber JE. TBCRC 031: Randomized Phase II Study of Neoadjuvant Cisplatin Versus Doxorubicin-Cyclophosphamide in Germline BRCA Carriers With HER2-Negative Breast Cancer (the INFORM trial). J Clin Oncol. 2020 May 10;38(14):1539-1548. doi: 10.1200/JCO.19.03292. Epub 2020 Feb 25. PMID 32097092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 13 academic centers and participants were recruited from these locations. Accrual occurred between January 2012 and January 2019.
Period: Overall Study
Arm/Group | Doxorubicin-Cyclophosphamide | Cisplatin
Started | 58 | 60
Completed (Participants received allocated intervention) | 57 (1 patient withdrew after 3 cycles; 5 patients received additional non-protocol chemo before surgery) | 60 (4 pts received <4 cycles of assigned chemo; 2 pts received add'l non-protocol chemo before surgery)
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxorubicin-Cyclophosphamide | Cisplatin | Total
Number analyzed (Participants) | 58 | 60 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (10) | 40 (9) | 42 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 117
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 49 | 48 | 97
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 44 | 43 | 87
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 5 | 5 | 10
BRCA status [Count of Participants; unit: Participants] — Eligible patients had a germline pathogenic or likely pathogenic variant (i.e. mutation) in BRCA1 or BRCA2; genetic testing was not performed as part of the trial, but known genetic status was required for eligibility
  Participants
    BRCA 1 | 37 | 44 | 81
    BRCA 2 | 20 | 15 | 35
    BRCA 1 and BRCA 2 | 1 | 1 | 2
Tumor size by imaging [Median (Inter-Quartile Range); unit: centimeters] | 2 [2 to 4] | 3 [2 to 4] | 2 [2 to 4]
T Stage (Tumor Size) [Count of Participants; unit: Participants] — Per National Cancer Institute (NCI) definition, T describes the size of the tumor and any spread of cancer into nearby tissue. The higher the T number, the larger the tumor and/or the more it has grown into nearby tissues.
  T1: The tumor in the breast is 20 millimeters (mm) or smaller in size at its widest area.
  T2: The tumor is larger than 20 mm but not larger than 50 mm.
  T3: The tumor is larger than 50 mm.
  Participants
    T1 | 17 | 12 | 29
    T2 | 31 | 35 | 66
    T3 | 10 | 12 | 22
    unknown | 0 | 1 | 1
N stage [Count of Participants; unit: Participants] — Per the National Cancer Institute Definition: N stage refers to the number of nearby lymph nodes that have cancer.
  N0: There is no cancer in nearby lymph nodes. N1, N2, N3: Refers to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer.
  Participants
    N0 | 34 | 31 | 65
    N1 | 19 | 24 | 43
    N2 | 2 | 2 | 4
    N3 | 3 | 3 | 6
Node status: biopsy before chemotherapy [Count of Participants; unit: Participants]
  positive | 24 | 29 | 53
  negative | 34 | 31 | 65
Stage [Count of Participants; unit: Participants] — Per the National Cancer Institute Definitions:
  Stage of Cancer.
  For Stage I, II, III, cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Participants
    I | 15 | 8 | 23
    II | 34 | 40 | 74
    III | 9 | 12 | 21
Estrogen Receptor (ER) [Count of Participants; unit: Participants]
  Positive (>/= 1%) | 20 | 20 | 40
  Negative (< 1%) | 38 | 40 | 78
Hormone receptor 1% cutoff [Count of Participants; unit: Participants] — ER= estrogen receptor; PR= progesterone receptor
  Participants
    Triple Negative Breast Cancer (ER & PR < 1%) | 36 | 40 | 76
    ER+ or PR+ | 22 | 20 | 42
Histology [Count of Participants; unit: Participants]
  Invasive ductal | 52 | 57 | 109
  Invasive lobular | 2 | 2 | 4
  Mixed | 3 | 1 | 4
  Other | 1 | 0 | 1
Pre-chemotherapy tumor grade [Count of Participants; unit: Participants] — Per the National Cancer Institute Definition: Tumor grade is description of tumor based on how abnormal the tumor cells and tumor tissue look under a microscope.
  In general, tumors are graded as 1, 2, 3, or 4, depending on the amount of abnormality. In Grade 1 tumors, the tumor cells and organization of the tumor tissue appear close to normal. These tumors tend to grow and spread slowly. In contrast, the cells and tissue of Grade 3 and Grade 4 tumors do not look like normal cells and tissue. Grade 3 and Grade 4 tumors tend to grow rapidly and spread faster than tumors with a lower grade.
  Participants
    1 | 1 | 2 | 3
    2 | 12 | 11 | 23
    3 | 45 | 46 | 91
    unknown | 0 | 1 | 1
Lymphovascular invasion [Count of Participants; unit: Participants]
  Present | 11 | 12 | 23
  Absent | 47 | 48 | 95
lymphocytic infiltrate [Count of Participants; unit: Participants]
  moderate/marked | 22 | 21 | 43
  absent/scant | 33 | 36 | 69
  unknown | 3 | 3 | 6
Stromal TILs [Median (Inter-Quartile Range); unit: percentage of stromal TILs] — TILs= tumor infiltrating lymphocytes
  The pre-chemotherapy clinical biopsy was assessed for tumor infiltrating lymphocytes. Population: Stromal TILS missing for 5 in Doxorubicin-Cyclophosphamide arm and 4 in the Cisplatin arm
  percentage of stromal TILs
    number analyzed (Participants) | 53 | 56 | 109
    (all) | 10 [1 to 20] | 10 [3 to 30] | 10 [1 to 20]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Pathologic Complete Response (pCR)
Description: Pathologic complete response (pCR) rate (determined by the Miller-Payne method) in doxorubicin-cyclophosphamide vs cisplatin arms.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin-Cyclophosphamide | Cisplatin
Number analyzed (Participants) | 57 | 60
Participants | 0 | 0
Statistical Analysis 1: Comparison: Doxorubicin-Cyclophosphamide vs Cisplatin; Test type: Other; Risk Ratio (RR) = .70, 90% CI 2-sided [0.39 to 1.2] — The risk ratio is comparing cisplatin to doxorubicin-cyclophosphamide (AC)

2. Secondary Outcome: Rate of Residual Cancer Burden (RCB) 0/1
Description: Residual Cancer Burden (RCB) rate of RCB 0 or 1 in participants receiving Doxorubicin-Cyclophosphamide vs participants receiving Cisplatin.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Doxorubicin-Cyclophosphamide | Cisplatin
Number analyzed (Participants) | 57 | 60
percentage of participants | 46 | 33
Statistical Analysis 1: Comparison: Doxorubicin-Cyclophosphamide vs Cisplatin; Test type: Other; Risk Ratio (RR) = .73, 90% CI 2-sided [.5 to 1.1] — The risk ratio is comparing cisplatin to doxorubicin-cyclophosphamide (AC)

3. Secondary Outcome: Clinical Response Rate
Description: Clinical response rate, defined as the number of partial and complete responses, after preoperative therapy with either cisplatin or AC in participants with germline BRCA mutation and breast cancer.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI or ultrasound: Complete Response (CR) = Disappearance of all target lesions; Partial Response (PR) is >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin-Cyclophosphamide | Cisplatin
Number analyzed (Participants) | 58 | 60
Participants | 43 | 45

4. Secondary Outcome: Number of Grade 3 and Grade 4 Adverse Events
Description: Comparison of toxicities for cisplatin and AC preoperative chemotherapy in BRCA mutation carriers with newly diagnosed breast cancer, reported as number of all Grade 3 and 4 adverse events and number of non-hematologic Grade 3 and 4 adverse events.
Time Frame: 2 years
Measure: Number; unit: Adverse Events
Arm/Group | Doxorubicin-Cyclophosphamide | Cisplatin
Number analyzed (Participants) | 57 | 60
Adverse Events
  All Grade 3 & 4 Adverse Events | 15 | 16
  Non-hematologic Grade 3 & 4 Adverse Events | 4 | 11

5. Secondary Outcome: Analysis of Pre-chemotherapy Biopsies
Description: Biopsies collected for future analyses of biomarkers that predict for response to cisplatin or AC chemotherapy in BRCA mutation carriers. Pretreatment tumor biopsies will be analyzed using genome wide SNP profiling to determine number of regions of telomeric allelic imbalance (NtAI) and chromosome 15q26 copy number, and chromosome 8q22 copy number. Tumor sections will be examined for gene amplifications, losses and NtAI in tumors. Gene expression profiling will be performed to determine intrinsic subtype (basal-like, claudin-low, etc.) and to measure biomarker genes including BLM and FANCI associated with cisplatin sensitivity or LAPTM4B and YWHAZ associated with anthracycline resistance. Exploratory analysis will be performed to seek new measures of therapy response using the data from DNA copy number and gene expression profiles. In addition, we will plan to perform whole exome and possibly whole genome sequencing of tumors to identify potential modifiers of response to therapy.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2025-08

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from time of treatment start, during treatment, and until 30 days after the last dose of treatment, about 3 months on average per participant, an average of 2 years.
Arm/Group | Doxorubicin-Cyclophosphamide | Cisplatin
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/60
Serious Adverse Events (participants affected / at risk) | 6/57 | 5/60
Other Adverse Events (participants affected / at risk) | 55/57 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin-Cyclophosphamide (N=57) | Cisplatin (N=60)
Allergic Reaction (Immune system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 2
Breast Infection (Infections and infestations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 4 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Increased Creatinine (Investigations) | 0 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin-Cyclophosphamide (N=57) | Cisplatin (N=60)
Fatigue (General disorders) | 45 | 48
Nausea (Gastrointestinal disorders) | 40 | 52
Tinnitus (Ear and labyrinth disorders) | 0 | 32
Vomiting (Gastrointestinal disorders) | 9 | 13
Diarrhea (Gastrointestinal disorders) | 10 | 7
Decreased Neutrophil Count (Investigations) | 5 | 8
Decreased White Blood Cell Count (Investigations) | 5 | 4
Decreased lymphocyte count (Investigations) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 31 | 4 — Note: Hair loss could not be accurately assessed for patients receiving AC, since hair loss was anticipated in this study before initiation of scalp cooling techniques and many patients shaved their hair in anticipation.
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3
Headache (Nervous system disorders) | 7 | 4
Constipation (Gastrointestinal disorders) | 20 | 13
Anemia (Blood and lymphatic system disorders) | 13 | 15
Oral Mucositis (Gastrointestinal disorders) | 15 | 7
Dysgeusia (Nervous system disorders) | 14 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT01670500/Prot_SAP_000.pdf